CLINICAL TRIAL: NCT06680661
Title: ABBA CORD: Double Umbilical Cord Blood Transplants With Abatacept for Graft Versus Host Disease Prophylaxis
Brief Title: ABBA CORD: dCBT w/ Abatacept for aGVHD Prophylaxis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Leland Metheny (Other)
Responsible Party: Sponsor-Investigator, Leland Metheny, Dr. Leland Metheny, Case Comprehensive Cancer Center
Organization: Case Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE1924
Record Dates: First submitted 2024-10-31; First posted 2024-11-08 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Acute Myelogenous Leukemia; Acute Lymphatic Leukemia; Chronic Myelogenous Leukemia; Myelodysplastic Syndromes; Myelodysplastic Syndrome Other; Chronic Myelomonocytic Leukemia; Lymphoma; Hodgkin Lymphoma
Keywords: Chronic Myelomonocytic Lymphoma; Umbilical Cord Blood Transplant; Double Umbilical Cord Transplant; Cord blood
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic; Lymphoma; Hodgkin Disease | interventions — Cyclophosphamide; fludarabine; Thiotepa; Whole-Body Irradiation; Tacrolimus; Mycophenolic Acid; Abatacept

STUDY DESIGN:
Intervention Model Description: Approximately 20 subjects will be enrolled in this trial: 7 patients will be accrued for the Stage 1. Stage 1 must be complete and the 7th patient reach T+180 prior to enrolling 13 additional patients to Stage 2.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cy/Flu/Thio/TBI + dCBT + Tac/MMF + Abatacept (Experimental): Cyclophosphamide (Cy), fludarabine (Flu), thiotepa (Thio), and total body irradiation (TBI) is the preparative regimen for Double Umbilical Cord Transplant (dCBT).
  Graft-versus-host disease prophylaxis will consist of tacrolimus (Tac) and mycophenolate mofetil (MMF). Abatacept will be administered.
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Thiotepa; Radiation: Total Body Irradiation; Biological: Double Umbilical Cord Transplant; Drug: Tacrolimus; Drug: Mycophenolate Mofetil; Drug: Abatacept

INTERVENTIONS:
Drug: Cyclophosphamide — Cyclophosphamide (Cy) is one part of the conditioning regimen. 50 mg/kg beginning on day -6.
Drug: Fludarabine — Fludarabine (Flu) is one part of the conditioning regimen. 150 mg/m2 (30 mg/m2 per day on days -6 to -2)
Drug: Thiotepa — Thiotepa (Thio) is one part of the conditioning regimen.10 mg/kg (5 mg/kg per day on days -5 and -4)
Radiation: Total Body Irradiation — 400 cGy (200 cGy per day on days -2 and -1).
Biological: Double Umbilical Cord Transplant — Cord blood is a regulated biologic. Selection of cord blood units will be based on published guidelines.
Drug: Tacrolimus — Tacrolimus will be administered post transplant. Graft-versus-host disease prophylaxis will consist of tacrolimus and mycophenolate mofetil (MMF), starting on day-5. Tacrolimus will continue at least until day 180 and then be tapered off.
Drug: Mycophenolate Mofetil — MMF will be administered post transplant. Graft-versus-host disease prophylaxis will consist of tacrolimus and mycophenolate mofetil (MMF), starting on day-5. MMF will continue until day 30.
Drug: Abatacept — Abatacept at a dose of 10mg/kg will be given on days T-1, T+5, T+14 and T+28.

SUMMARY:
The goal of this clinical trial is to see if adding abatacept to tacrolimus and MMF prevents or reduces the chances of acute graft versus host disease which is a complication that can occur after transplant in participants with blood cancer. The usual therapy for graft versus host disease prevention after a cord blood transplant includes tacrolimus and MMF. The main question this clinical trial aims to answer is whether or not abatacept will be safe and effective in reducing aGVHD rates in dCBT.

Participants will:

* Partake in exams, tests, and procedures as part of usual cancer care.
* Partake in conditioning, which is the treatment that is given before a transplant.
* Have a cord blood transplant.
* Partake in radiation following the transplant.

DETAILED DESCRIPTION:
Cord blood (CB) is a valuable alternative graft source for patients with hematologic malignancies in need of allogeneic transplantation who lack human leukocyte antigen (HLA)-matched adult donors. In Black, Asian, Hispanic populations, the chance of finding a HLA matched donor is 23%, 41%, and 46%, respectively. CB allows for greater HLA difference between donor and recipient, and increases the availability of donors, and therefore transplant, to these populations. Retrospective analyses and prospective trials demonstrate that recipients of double CB transplant (dCBT) have a grade II-IV acute graft versus host disease (aGVHD) rate of 45-90% and grade III-IV aGVHD rates up to 24%. This high aGVHD rate is likely due to the HLA-disparities between donor and recipient, which also drives a robust graft versus leukemia response8. Anti-thymocyte globin has been used in dCBT to reduce the incidence of aGVHD, but is no longer recommended due to delayed immune-reconstitution of the CB grafts. The ABA2 trial demonstrated efficacy and safety of abatacept as prophylaxis for aGVHD in HLA-mismatched unrelated donors (MMUD), significantly reducing the rate both of grade III-IV aGVHD and grade II-IV aGVHD in 7/8 MMUD when compared to historical controls. Our hypothesis is that abatacept will be safe and effective in reducing aGVHD rates in dCBT.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the following hematologic malignancies:

  * Acute myelogenous leukemia (AML): High-risk and intermediate-risk AML including:

    * Antecedent hematological disease (e.g., myelodysplasia (MDS))
    * Treatment-related leukemia
    * Complete Remission (CR1) with poor or intermediate-risk cytogenetics or molecular markers (e.g. Flt 3 mutation, 11q23, del 5, del 7, complex cytogenetics)
    * CR2 or CR3
    * Induction failure or 1st relapse with < 10% blasts in the marrow
  * Acute lymphoblastic leukemia (ALL):

    * High-risk CR1 including:

      * Poor-risk cytogenetics (e.g., Philadelphia chromosome t(9;22)or 11q23 rearrangements)
      * Philadelphia chromosome-like ALL
      * Presence of minimal disease by flow cytometry after 2 or more cycles of chemotherapy
    * No CR within 4 weeks of initial treatment
    * Induction failure with < 10% blasts in the marrow
    * CR2 or CR3
  * Myelodysplastic syndromes (MDS), Intermediate, High or Very High Risk by the revised international prognostic scoring system or treatment related MDS.
  * Bi-phenotypic or mixed-phenotypic acute leukemia in:

    * CR.
    * Induction failure or 1st relapse with < 10% blasts in the marrow.
  * Chronic Myelogenous Leukemia (CML) in second chronic phase after accelerated or blast crisis.
  * Chronic Myelomonocytic Leukemia (CMML)
  * Hodgkin's Lymphoma that is relapsed or refractory
* Age > or equal to 18 years, < or equal to 70yrs
* KPS > or equal to 80 for Flu/Cy/Thio/TBI; KPS > 60 for Flu/Treo/TBI
* Patients without a suitable HLA-matched related or unrelated donor
* Patient with the following CB units:

  * At least two 4-8/8 HLA high resolution matched CB units. Both must have a cell dose of 1.5x107 TNC/kg each and 1.5x105 CD34+/kg
  * A minimum of 1 CB unit as back up.
* Concurrent Therapy for Extramedullary Leukemia or CNS Lymphoma: Concurrent therapy or prophylaxis for testicular leukemia, CNS leukemia, and CNS lymphoma including standard intrathecal chemotherapy and/or radiation therapy will be allowed as clinically indicated. Such treatment may continue until the planned course is completed. Subjects must be in CNS remission at the time of protocol enrollment if there is a history of CNS involvement. Maintenance therapy after transplant is allowed.
* Subjects must have the ability to understand and the willingness to sign a written informed consent document.
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use a contraceptive method with a failure rate of < 1% per year during the treatment period and for 12 months after the last dose of abatacept.
* A woman is considered to be of childbearing potential if she is < 60 years old, postmenarcheal, has not reached a postmenopausal state (< 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus).

  * Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices.

The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.

* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures with female partners of reproductive potential, and agreement to refrain from donating sperm, as defined below:

  * With female partners of childbearing potential, men must remain abstinent or use a condom plus an additional contraceptive method that together result in a failure rate of < 1% per year during the treatment period and for 12 months after the last dose of abatacept. Men must refrain from donating sperm during this same period. With pregnant female partners, men must remain abstinent or use a condom during the treatment period and for at least 12 months after the last dose of abatacept.
  * The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.

Exclusion Criteria:

* Patients with inadequate Organ Function as defined by:

  * Creatinine clearance < 50ml/min
  * Bilirubin > 2X institutional upper limit of normal unless Gilbert syndrome
  * AST (SGOT) > 3X institutional upper limit of normal
  * ALT (SGPT) > 3X institutional upper limit of normal
  * Pulmonary function: DLCOc < 60% normal
  * Cardiac: left ventricular ejection fraction < 50
* Patients with uncontrolled inter-current illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant or breastfeeding women are excluded from this study because chemotherapy involved with RIC have the significant potential for teratogenic or abortifacient effects.
* Any condition that would, in the investigator's judgment, interfere with full participation in the study, including administration of study drug and attending required study visits; pose a significant risk to the subject; or interfere with interpretation of study data.
* Known allergies, hypersensitivity, or intolerance to any of the study medications, excipients, or similar compounds.
* Presence of donor-specific antibodies against chosen graft source.
* Hematopoietic Cell Transplantation Comorbidity index (HCT-CI) > 5.
* Prior autologous or allogenic stem cell transplant within the preceding 12 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-02-25 (Actual); Primary Completion 2027-10-29 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
Severe aGVHD free survival | 180 days after treatment
  To assess severe aGVHD (grade III-IV acute GVHD) free survival (SGFS) at T+180.

SECONDARY OUTCOMES:
Non-relapse mortality | 1 year post transplant
  Treatment Related Mortality (TRM) at 1 year is the percentage of patients who expire from treatment related toxicity attributed to transplant up to 1 year after transplant.
Overall Survival | 1 year post transplant
  Overall Survival (OS) at 1 year is the percentage of patients alive at 1 year after transplant.
Rate of relapse | 1 year post transplant
  Relapse incidence at 1 year is the percentage of patients who experience relapse of their hematologic malignancy up to 1 year after transplant.
Disease free survival | 1 year post transplant
  Disease Free Survival at 1 year is the percentage of patients alive and without evidence of hematologic malignancy at 1 year after transplant.
Incidence of chronic GVHD | 1 year post transplant
  Chronic graft versus host disease (cGVHD) 1-year cumulative incidence is the percentage of patients who experienced any cGVHD up to 1 year after transplant.
Incidence of chronic GVHD | 2 years post transplant
  Chronic graft versus host disease (cGVHD) 2-year cumulative incidence is the percentage of patients who experienced any cGVHD up to 2 years after transplant.
Incidence of chronic GVHD | 3 years post transplant
  Chronic graft versus host disease (cGVHD) 3-year cumulative incidence is the percentage of patients who experienced any cGVHD up to 3 years after transplant.
Rate of Grade III-IV aGVHD | 100 days after treatment
  Grade III-IV aGVHD prevalence at T+100 is the percentage of patients who have grade III-IV aGVHD at T+100.
Rate of Grade II-IV aGVHD | 100 days after treatment
  Grade II-IV aGVHD prevenance at T+100 is the percentage of patients who have grade II-IV aGVHD at T+100.
Rate of Grade III-IV aGVHD | 180 days after treatment
  Grade III-IV aGVHD prevalence at T+180 is the percentage of patients who have grade III-IV aGVHD at T+180.
Rate of Grade II-IV aGVHD | 180 days after treatment
  Grade II-IV aGVHD prevalence at T+180 is the percentage of patients who have grade II-IV aGVHD at T+180.
CMV reactivation rate | 1 year after transplant
  The cumulative incidence of CMV reactivation at 1 year is defined as the detection of CMV within any organ by biopsy or within the plasma within the first year of transplant.
EBV reactivation rate | 1 year after treatment
  The cumulative incidence of EBV reactivation at 1 year is defined as the detection of EBV in the plasma or blood less than 1000 copies/ml within the first year of transplant.
Time to neutrophil engraftment | Within first 30 days of transplant
  Neutrophil engraftment will be calculated as the days from transplant where the absolute neutrophil count (ANC) reaches >500cells/ul x 3 days.
Time to platelet engraftment | Within first 60 days of transplant
  Platelet engraftment will be calculated as the days from transplant where the platelet count reaches 20,000 platelets /ul without the need of transfusion of platelets for 7 days.
Donor chimerism | Day 100 post transplant
  Donor chimerism rates will drawn at day 100 post transplant.
Donor chimerism | 1 year post transplant
  Donor chimerism rates will drawn 1 year post transplant.
Time to taper off tacrolimus | Within 1 year of transplant
  The average time to taper off of tacrolimus will be calculated.
Time to taper off MMF | Within 90 days of transplant
  The average time to taper off of mycophenolate mofetil (MMF) will be calculated.
Assessment of aGVHD biomarker ST2 | 7 days post transplant
  An assessment of aGVHD biomarker ST2 will occur 7 days post transplant.
Assessment of aGVHD biomarker ST2 | 28 days post transplant
  An assessment of aGVHD biomarker ST2 will occur 28 days post-transplant.
Assessment of aGVHD biomarker REG3α | 7 days post transplant
  An assessment of aGVHD biomarker REG3α will occur 7 days post-transplant.
Assessment of aGVHD biomarker REG3α | 28 days post transplant
  An assessment of aGVHD biomarker REG3α will occur 28 days post-transplant.

CONTACTS AND LOCATIONS:
Overall Officials: Leland Metheny, MD, Principal Investigator — University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (1):
- University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in publication.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Compiled and analyzed patient data will be published upon study completion. Publisher may request Protocol and Statistical Analysis Plan.